CLINICAL TRIAL: NCT02900703
Title: Epidemiological Surveillance of Rotavirus Gastroenteritis With a Perspective of Vaccination
Brief Title: Surveillance of Rotavirus Gastroenteritis
Acronym: Rotavirus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: POTHIER Sanofi 2011
Record Dates: First submitted 2016-09-05; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- PATIENT
  Interventions: Biological: stool samples

INTERVENTIONS:
Biological: stool samples

SUMMARY:
* Epidemiological studies have shown the diversity of resistance genotypes and the evolution of their prevalence in the paediatric population. This large study conducted in a context of very low vaccination coverage will generate more precise data on the natural epidemiological evolution of rotavirus, notably the G9 genotype, which has appeared relatively recently.
* This study will allow us to identify and document rare or unusual strains of human or animal origin. The complete genetic characterization of these strains will also make it possible to study their ability to recombine and to assess the risk of emergence. Among these still rare strains, the investigators are particularly monitoring G12 rotavirus, whose ability to recombine raises the risk of emergence.
* For at least one of the centres taking part in the study, the paediatric population studied will be given strong vaccination coverage. It will be extremely interesting to compare the results obtained in the vaccinated population with non-vaccinated children to assess the impact of this vaccination on the distribution of rotavirus genotypes

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized or consulting in one of the participating centres since January 2007 for acute gastroenteritis (AGE). AGE is defined by at least 3 soft or liquid stools or at least 3 bouts of vomiting within 24 hours or one of the following signs - diarrhoea or vomiting accompanied by at least 2 additional symptoms among diarrhoea or vomistin, abdominal pain, fever.

Exclusion Criteria:

* Children older than 5 years.
* Children presenting chronic diarrhoea (> 2 weeks).
* Children presentant immune deficiency.
* Children presenting nosocomial gastroenteritis. The nosocomial nature will be determined by the onset of acute diarrhoea occuring after 48 hours following admission

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children presenting gastroenteritis
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2007-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
number of viral strains of rotavirus | through the completion study an average 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France